CLINICAL TRIAL: NCT01421082
Title: Evaluation of Physiologic Parameters to Study the Mechanism of Action of the PneumRx, Inc. Lung Volume Reduction Coil (LVRC) in Subjects With Homogeneous Emphysema
Brief Title: Evaluation of Physiologic Parameters to Study the Mechanism of Action of the Lung Volume Reduction Coil in Subjects With Homogeneous Emphysema
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: PneumRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN0012
Record Dates: First submitted 2011-08-18; First posted 2011-08-22 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Emphysema
Keywords: LVRS (Lung Volume Reduction Surgery); LVRC (Lung Volume Reduction Coil); Emphysema; coil; RePneu
MeSH Terms: conditions — Emphysema | interventions — Pneumonectomy; Anterior Temporal Lobectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LVRC Treatment (Experimental)
  Interventions: Device: Lung Volume Reduction Coil (LVRC) (PneumRx, Inc.)

INTERVENTIONS:
Device: Lung Volume Reduction Coil (LVRC) (PneumRx, Inc.) — Lung Volume Reduction Coil (LVRC)
  Other Names: Lung Volume Reduction Surgery (LVRS); Lobectomy

SUMMARY:
The PneumRx Lung Volume Reduction Coil (LVRC) has been shown to effectively improve quality of life, exercise capacity, and static lung volumes, in patients with emphysema. The mechanism of action for these effects is believed to be related to the restoration of elastic recoil to lung parenchyma that has been damaged by emphysema. The objective of this study is to evaluate several physiologic parameters which should provide measures directly related to the mechanism of action by which the coils produce these outcomes.

ELIGIBILITY:
Inclusion Criteria:

Subject > 35 years of age CT scan indicates homogeneous emphysema Subject has stopped smoking for a minimum of 6 months prior Subject (and legal guardian if applicable) read, understood and signed the Informed Consent form

Exclusion Criteria:

Subject has a history of recurrent clinically significant respiratory infection Subject has uncontrolled pulmonary hypertension Subject has evidence of other disease that may compromise survival such as lung cancer, renal failure, etc Subject is pregnant or lactating Subject has an inability to tolerate bronchoscopy Subject has clinically significant bronchiectasis Subject has giant bullae Subject has had previous LVR surgery, lung transplant or lobectomy Subject has been involved in other pulmonary drug studies with 30 days prior Subject has other condition that would interfere with completion of study, follow up assessments or that would adversely affect outcomes

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
6 minute walk test (6MWT) | 6 months
  The primary effectiveness endpoint will be the improvement in the 6 minute walk test (6MWT) from Baseline compared to Follow-Up.

SECONDARY OUTCOMES:
Adverse Events | 6 months
  The safety objective of this study is to identify the adverse effects attributed to device.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen - UMCG, Groningen, The Netherlands, Netherlands